CLINICAL TRIAL: NCT07350629
Title: A Study on Noninvasive Real-Time Arterial Pressure Waveform Analysis for the Detection and Evaluation of Cardiovascular Diseases
Brief Title: Noninvasive Real-Time Arterial Waveform Monitoring for Cardiovascular Disease Assessment
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaojing, Chief Physician, Anhui Provincial Cancer Hospital
Other Study IDs: 2025-APW-001
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Aortic Regurgitation Disease; Aortic Stenosis Disease; Healthy Subjects

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Subjects: Healthy adult volunteers with no known cardiovascular disease will undergo noninvasive arterial waveform acquisition using the photoacoustic imaging device. No intervention is applied; data collection provides baseline waveform features for comparison with AR and AS patients.
- Aortic Regurgitation (AR) Patients: Participants diagnosed with aortic regurgitation (AR) will undergo noninvasive arterial waveform acquisition using a photoacoustic imaging device. No intervention is applied; data collection focuses on capturing finger arterial pulse waveforms to assess features associated with AR.
- Aortic Stenosis (AS) Patients: Participants diagnosed with aortic stenosis (AS) will undergo noninvasive arterial waveform acquisition using the same photoacoustic imaging device. No intervention is applied; data collection focuses on capturing finger arterial pulse waveforms to assess features associated with AS.

SUMMARY:
The goal of this observational study is to learn whether noninvasive real-time arterial waveform monitoring can be used to assess cardiovascular diseases in adults. The main question it aims to answer is:

Can photoacoustic imaging accurately capture arterial waveforms from patients' fingers? Can features extracted from the arterial waveforms reflect the type and severity of cardiovascular diseases? Participants will be asked to place their fingers into the imaging device, where their finger arterial pulse information will be noninvasively recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Able to provide informed consent
* For AR group: clinically diagnosed aortic regurgitation
* For AS group: clinically diagnosed aortic stenosis
* For healthy controls: no history of cardiovascular disease
* Able to undergo finger arterial waveform measurement

Exclusion Criteria:

* History of recent cardiac surgery or intervention (<6 months)
* Hand disorders affecting finger mobility (e.g., arthritis)
* Pregnant or breastfeeding women
* Participation in other studies affecting arterial waveform
* Unable to understand or comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from adult patients attending the cardiology department at the First Affiliated Hospital of University of Science and Technology of China, including individuals diagnosed with aortic regurgitation (AR) or aortic stenosis (AS), as well as healthy adult volunteers without known cardiovascular disease. Recruitment will focus on adults aged 18-80 years who are able to comply with finger arterial waveform measurement procedures.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the state of aortic regurgitation and aortic stenosis by photoacoustic tomography | At enrollment (single time point)
  To determine the feasibility of using photoacoustic tomography to differentiate aortic regurgitation and aortic stenosis based on arterial waveform measurements.

SECONDARY OUTCOMES:
Rise time of photoaocustic arterial waveform | At enrollment (single time point)
  To determine the systolic upstroke rise time of arterial waveforms using photoacoustic tomography
Decay time of photoaocustic arterial waveform | At enrollment (single time point)
  To determine the diastolic decay time of arterial waveforms using photoacoustic tomography
Dicrotic notch time of photoaocustic arterial waveform | At enrollment (single time point)
  To determine the dicrotic notch time of arterial waveforms using photoacoustic tomography

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China